CLINICAL TRIAL: NCT05131763
Title: A Phase I Clinical Trial of NKG2D-based CAR T-cells Injection for Subjects With Relapsed/Refractory NKG2DL+ Solid Tumors
Brief Title: NKG2D-based CAR T-cells Immunotherapy for Patient With r/r NKG2DL+ Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: KAEDI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan-Changchun
Record Dates: First submitted 2021-11-05; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma; Glioblastoma; Medulloblastoma; Colon Cancer
Keywords: NKG2D-based CAR T-cells; solid tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Glioblastoma; Medulloblastoma; Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD-025 (Experimental): NKG2D-based CAR T-cells Injection; Dosage:1-10x10^6/kg, 70ml/time, The CAR-T cells will be administered by i.v. or hepatic portal artery injection over 20-30 minutes Frequency: total one time
  Interventions: Biological: NKG2D-based CAR T-cells

INTERVENTIONS:
Biological: NKG2D-based CAR T-cells — Autologous genetically modified anti-NKG2DLs CAR transduced T cells

SUMMARY:
The primary objective of this study is to evaluate the safety and clinical activity of NKG2D-based CAR-T cells infusion in the treatment of relapsed/refractory NKG2DL+ solid tumors.

DETAILED DESCRIPTION:
The preclinical study clarified that NKG2D-based CAR-T cells showed strong cytotoxicity against NKG2DL+ cell lines in vitro as well as a therapeutic effect against NKG2DL+ cell xenografts in vivo. In addition, the data also demonstrated the safety of NKG2D-based CAR-T therapy. NKG2D-based CART represent a potentially effective and safety therapeutic approach for patient with relapsed/refractory NKG2DL+ solid tumors. In this trial, the investigators researched the safety of administering NKG2D-based CAR-T which generated with CD8 hinge region and transmembrane region, 4-1BB costimulatory region and CD3 zeta region. The investigators also assessed that disease response was determined within the context of a phase I trial.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women≥18 years old,
2. Patient with NKG2DL+ cell tumors confirmed by pathology and histology,
3. Fail or unwilling to receive first-line treatment,
4. Disease must be measurable according to the corresponding guidelines,
5. Main organs function normally and meet following requirements:

   Routine blood index#No Blood transfusion within 14 days# 1)HB≥90g/ L; 2)ANC≥1.5×109/L; 3)PLT≥75×109/L# Serum biochemicals index 1) BIL <1.5 upper normal limit (ULN); 2) ALT and AST<2.5×ULN; In the case of liver metastasis, ALT and AST<5×ULN; 3) Serum Cr≤1×ULN, endogenous creatinine clearance≥50ml/min (Cockcroft-Gault formula); 4) ECOG physical condition score: 0-2
6. Expected survival time ≥3 months,
7. Patient with adequate bone marrow reserve, hepatic and renal functions,
8. No other uncontrolled diseases such as lung, kidney and liver infection before enrollment,
9. Women of child-bearing age must undergo a negative pregnancy test (serum or urine) within 7 days prior to enrollment and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last dose; men should agree to contraception during the observation period and within 8 weeks of the last dose,
10. Patients voluntarily participated in this trial and sign the informed consent form,
11. Patients with compliance and expected to follow up the efficacy and adverse reactions as required by the protocol,

Exclusion Criteria:

* 1. Pregnant or lactating women, 2. Patients who need to use systemic steroids at the same time, 3. Under following treatment conditions currently: 1) during the other antitumor clinical observation period within 14 days before blood collection; 2) patient has not recovered from acute side effects of the previous treatment; 4. Receive radiotherapy within 4 weeks before enrollment, 5. Patients who received any other cell therapy before, 6. Patients with unqualified T cell amplification efficiency, 7. Uncontrolled symptoms or other illnesses, including but not limited to infection, congestive heart failure, unstable angina, arrhythmia, psychosis, 8. Patients with severe acute allergic reactions, 9. Patients who have received other cell therapies, 10. Other serious conditions that may limit patient's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 3 months.
  The number of patiens who suffered ≥ 3 grade toxicities according to the CTCAE criteria after CAR-T therapy.
Detailed adverse events post NKG2D-based CAR-T therapy. | through study completion, an average of 3 months.
  The events included infusion reactions, CRS, tumor lysis syndrome and hematological toxicity. The criteria mainly reffered to guidelines for immune related adverse reactions.

SECONDARY OUTCOMES:
overall survival (OS) | 2 years post infusion
  For all subjects, overall survival refers to the period from being included in the test group to death caused by any reason
Progress Free Survival (PFS) | 2 years post infusion
  Progress Free Survival after administration
Partial response rate | through study completion, an average of 3 months.
  According the RECISE 1.1 criteria, as to the measurable primary lesions, we measure the long and short diameter. As to unmeasurable primary leisons, we measure the measurable metastatic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: kuaile zhao, doctor, Study Director — Fudan University; Changchun Cai, doctor, Study Director — Xunyang Changchun Shihua Hospital
Locations (1):
- Xunyang Changchun Shihua Hospital, Jiujiang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No